CLINICAL TRIAL: NCT00911768
Title: PMS Clinical Study of Korean Red Ginseng Powder on Dry Mouth and Salivary Flow Rates in Xerostomatic Populations
Brief Title: Effect of Korean Red Ginseng (KRG) on Dry Mouth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Korean Society of Ginseng (Other)
Responsible Party: Jae-Woo Park, KMD, PhD, Kyung Hee East-West Neo Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2007-007
Record Dates: First submitted 2009-03-03; First posted 2009-06-02 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Xerostomia
Keywords: Xerostomia; Panax ginseng(Korean Red Ginseng); Visual Analogue Scale; Salivary Flow Rates
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Korean Red Ginseng group (Experimental): The brand name of experimental drug is 'Capsule of Korean Red Ginseng Powder'. It consists of the powder of steamed root of Panax ginseng made by Korean Ginseng Corp.
  Interventions: Dietary Supplement: Korean Red Ginseng Powder Capsule
- Corn-starch powder with ginseng flavor (Placebo Comparator): The placebo of this study is corn-starch powder with Korean Red Ginseng flavor. It has the same shape, color and flavor like experimental drug.
  Interventions: Dietary Supplement: Corn-starch powder with ginseng flavor

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng Powder Capsule — Generic name: Korean Red Ginseng Powder Capsule Original herb name: Panax ginseng Form and contents: Capsule with powder of steamed root of 6-year Panax ginseng Dosage and frequency: 6 g per day (twice a day), Oral administration Administration duration: 56 days in the study
  Other Names: Brand Name: Korean Red Ginseng Powder Capsule
  Arms: Korean Red Ginseng group
Dietary Supplement: Corn-starch powder with ginseng flavor — There is no specific name because this intervention is placebo. This placebo has the same form, color and flavor as Korean Red Ginseng Powder Capsule.
  The dosage form, dosage, frequency and duration is also same as experimental intervention (Korean Red Ginseng Powder Capsule).
  Main contents: corn-starch with Panax ginseng flavor
  Other Names: Corn-starch powder capsule with Korean Red Ginseng flavor
  Arms: Corn-starch powder with ginseng flavor

SUMMARY:
The purpose of this study is to determine the effect of KRG (Korean Red Ginseng) on Dry Mouth (Xerostomia).

DETAILED DESCRIPTION:
Korean Red Ginseng

* Worldwide use
* A main herb of old oriental prescriptions for dry mouth
* Need for correct information by RCT

ELIGIBILITY:
Inclusion Criteria:

* Dry mouth patients

Exclusion Criteria:

* Sjögren syndrome
* Irradiation related xerostomia
* Severe psychiatric diseases
* pregnancy or breast feeding women

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Woo Park, K.M.D., Ph.D, Principal Investigator — Kyung Hee East-West Neo Medical Center
Locations (1):
- Kyung Hee East-West Neo Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the waiting room and consulting room of Oriental Clinic of Gastrointestinal diseases and Chronic fatigue of Kyung Hee East-West Neo-Medical Center (Seoul, Korea) between September 2007 and February 2008
Pre-assignment Details: Totally, 133 participants were enrolled in the trial; 100 participants screened and 33 of them (women 18, men 15) were excluded because of abnormal liver function (1), present illness (2), a plan to pregnancy (1), and self refusals or disconnections (28).
Groups:
- Korean Red Ginseng: Capsules of Korean Red Ginseng Powder 3g administrated twice daily for 8 weeks.
- Placebo: Capsules of corn-starch powder with Korean Red Ginseng flavor 3g administrated twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Korean Red Ginseng | Placebo
Started | 50 | 50
Completed | 44 | 46
Not Completed | 6 | 4
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Korean Red Ginseng | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 44 | 45 | 89.0
  >=65 years | 6 | 5 | 11.0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.14 (15.97) | 46.02 (16.14) | 47.1 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54.0
  Male | 22 | 24 | 46.0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 50 | 50 | 100.0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale of Subjective Dry Mouth
Description: Visual Analogue Scale of Subjective Dry Mouth is 10 cm, where 0 cm indicates no dry mouth and 10 cm the severe dry mouth.
Time Frame: 8 weeks
Population: Because primay outcome of the study was changes of Visual Analogue Scale of Subjective Dry Mouth between 0, 4 and 8 weeks, per protocol analysis was applied.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Korean Red Ginseng | Placebo
Number analyzed (Participants) | 44 | 46
cm | 5.21 (2.02) | 5.03 (1.93)
Statistical Analysis 1: Comparison: Korean Red Ginseng vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.181, 95% CI [-0.647 to 1.008], Standard Error of Mean 0.416

2. Secondary Outcome: Stimulated Salivary Flow Rates
Description: Stimulated salivary flow rates were compared between 0 and 8 weeks in both groups.
Time Frame: 8 weeks
Population: Because secondary outcome of the study was also changes of stimulated salivary flow rates between 0 and 8 weeks, per protocol analysis was applied.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Korean Red Ginseng | Placebo
Number analyzed (Participants) | 44 | 46
ml/min | 1.046 (0.552) | 1.392 (0.549)
Statistical Analysis 1: Comparison: Korean Red Ginseng vs Placebo; Test type: Non-Inferiority or Equivalence — A non-inferiority analysis was conducted. We just compared the difference of stimulated salivary rates between both groups at 8 weeks, because there were no definition of the effective margin; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.346, 95% CI [-0.576 to -0.115], Standard Error of Mean 0.116

3. Secondary Outcome: Unstimulated Salivary Flow Rates
Description: Unstimulated salivary flow rates were compared between 0 and 8 weeks in both groups.
Time Frame: 8 weeks
Population: Because secondary outcome of the study was changes of unstimulated salivary flow rates between 0 and 8 weeks, per protocol analysis was applied.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Korean Red Ginseng | Placebo
Number analyzed (Participants) | 44 | 46
ml/min | 0.220 (0.153) | 0.266 (0.185)
Statistical Analysis 1: Comparison: Korean Red Ginseng vs Placebo; Test type: Non-Inferiority or Equivalence — A non-inferiority analysis was conducted. We just compared the difference of unstimulated salivary rates between both groups at 8 weeks, because there were no definition of the effective margin; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.086, 95% CI [-0.155 to -0.017], Standard Error of Mean 0.035

ADVERSE EVENTS:
Arm/Group | Korean Red Ginseng | Placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No